CLINICAL TRIAL: NCT04649671
Title: The Effect of Mobile Health-based Exercise on Insulin Sensitivity in Hepatocellular Carcinoma Patients With Insulin Resistance: A Randomized Controlled Trial
Brief Title: The Effect of Mobile Health-based Exercise on Hepatocellular Carcinoma Patients With Insulin Resistance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruitment and deficit of research fund
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Moon Seok Choi, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC2020-06-037
Record Dates: First submitted 2020-11-17; First posted 2020-12-02 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Hepatocellular Carcinoma; Insulin Resistance
MeSH Terms: conditions — Carcinoma, Hepatocellular; Insulin Resistance | interventions — Telemedicine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Hepatocellular carcinoma (HCC) patients with insulin resistance who underwent hepatic resection or radiofrequency ablation (RFA) will be enrolled. Patients included in the control arm will receive a booklet including information about physical activity recommendations and practice (education). After 12 weeks, they will also be provided mobile application and wearable device and perform exercise for 12 weeks.
- Mobile health (Active Comparator): HCC patients with insulin resistance who underwent hepatic resection or RFA will be enrolled. Patients included in the intervention arm will receive both booklet and mobile health program. They will perform exercise daily with mobile application and wearable device (warm-up, stretching, aerobic, and strengthening) for 24 weeks.
  Interventions: Behavioral: Mobile health

INTERVENTIONS:
Behavioral: Mobile health — Perform exercise daily with mobile application and wearable device (warm-up, stretching, aerobic, and strengthening).
  Mobile application: Hepatocellular carcinoma by Second Doctor Wearable device: Dofit
  Arms: Mobile health

SUMMARY:
Exercise is predicted to have positive effect among patients with hepatocellular carcinoma (HCC). However, little attention has been paid to the role of physical activity with wearable device in the management of HCC patients in the aspect of improvement in insulin resistance.

We designed this study to investigate whether personalized exercise with mobile health program improves insulin resistance without decompensation in HCC patients with insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 to 70 years
* Patients who were diagnosed with early-stage HCC, defined by modified UICC stage 1 or 2
* Patients with treatment-naive and recurrent HCC who have received treatment and achieved complete response at the time of screening
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Patients with insulin resistance (HOMA-IR >=2.2)

Exclusion Criteria:

* Child Pugh class B or C
* Alcohol intake >20g/day
* History of decompensation
* Severe medical comorbidities (ischemic heart disease, 3rd degree atrioventricular block, chronic obstructive pulmonary disease, severe hypertension (blood pressure > 200/120 mmHg) or psychiatric illnesses which limit ability to exercise safely
* Who takes insulin sensitizer (sulfonylurea, biguanide, thiazolidinedione, glucagon-like peptide-1 agonist, dipeptidyl peptidase-4 inhibitor) or uses insulin
* Uncontrolled diabetes mellitus (Hemoglobin A1c >10%)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Improvement of insulin resistance | After 12 weeks
  The proportion of normalization of homeostatic model assessment of insulin resistance (HOMA-IR) (<2.2)

SECONDARY OUTCOMES:
Improvement of insulin resistance | After 24 weeks
  The proportion of normalization of homeostatic model assessment of insulin resistance (HOMA-IR) (<2.2)
Improvement of 6-minute walk test | After 12 and 24 weeks
  - Changes in meters assessed using the 6-minute walk test
Improvement of grip strength test | After 12 and 24 weeks
  - Changes in kilograms assessed using grip strength test
Improvement of 30-second chair stand test | After 12 and 24 weeks
  - Changes in seconds assessed using 30-second chair stand test
Improvement of the score of International Physical Activity Questionnaire-Short Form (IPAQ-SF) | After 12 and 24 weeks
  - Changes in metabolic equivalents (METs) per week calculated using IPAQ-SF
Improvement of quality of life | After 12 and 24 weeks
  Improved score of European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire C30
Nutritional status | After 12 and 24 weeks
  Comparison of nutrition score using mini nutritional assessment
Adverse events | After 12 and 24 weeks
  Any adverse events occurred during exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Moon Seok Choi, Seoul, South Korea

REFERENCES:
- [Derived] Yeo SM, Oh JH, Yu HJ, Sinn DH, Hwang JH. The effect of mHealth-based exercise on Insulin Sensitivity for patients with Hepatocellular carcinoma and insulin resistance (mISH): protocol of a randomized controlled trial. Trials. 2022 Nov 8;23(1):930. doi: 10.1186/s13063-022-06858-w. PMID 36348422